CLINICAL TRIAL: NCT07041476
Title: HYBRID TELE-REHABILITATION VERSUS CLINIC-BASED THERAPY IN PATIENTS WITH LUMBAR RADICULOPATHY: A RANDOMIZED CONTROLLED TRIAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmed Adel Eid (Other)
Responsible Party: Sponsor-Investigator, Ahmed Adel Eid, Demonstrator, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 153488
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Lumbar Disc Prolapse With Radiculopathy
MeSH Terms: interventions — Exercise; Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HYBRID TELE-REHABILITATION (Experimental)
  Interventions: Other: Exercise; Other: telemedicine

INTERVENTIONS:
Other: Exercise — Tele-rehabilitation methods can provide an important advantage for patients who cannot receive hospital services due to pain, mobility limitations, and distance to the hospital
Other: telemedicine — Tele-rehabilitation will be achieved through a video conference (VC) via the internet platform Zoom at the time and day 29 decided upon with the therapist

SUMMARY:
A single blinded clinical randomized trial. A single blinded trained investigator examined all patients and collect all data to eliminate inter- investigator error. Patients will be divided according to the treatment procedure into two groups equal in numbers to investigate a comparative effect of hybrid tele-rehabilitation to clinic- based therapy in patients with lumbar radiculopathy.

ELIGIBILITY:
Inclusion Criteria:

-

1) Both genders will be involved, 2) Symptoms started within more than 4 weeks (Ghasabmahaleh et al., 2021). 3) Patients' age ranges from 25-45 years (Karthick et al., 2024). 4) All patients will be referred by the physician after confirmed diagnosis of lumbar radiculopathy at L4/5 or L5/S1 level through clinical assessment and imaging studies.

5) Patients have sufficient education level. 6) Body mass index for patients will be from 18.5 to 29.9.

Exclusion Criteria:

* 1) History of pelvic, hips, or spine surgery, 2) Any unstable lumbar condition such as spinal fractures, tumor, cauda equina syndrome and spondylolisthesis (Ghasabmahaleh et al., 2021).

History of neurological disorders causing radicular pain, 4) Any preexisting injury that may become exacerbated or made worse with participation (Zainab et al., 2022).

5) Cardiovascular problems (unstable angina, recent myocardial infarction within the last three months, congestive heart failure, significant heart valve dysfunction, or unstable hypertension) or pulmonary disorders (Vijayaraj., 2018).

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
numeric pain rating scale (NPRS) | 5 minutes
  The NPRS is frequently employed to measure pain intensity, in which patients are asked to select a number (from 0 to 10) to represent their pain severity before and after medical consultation
Oswestry disability index (ODI) | 5 minuets
  used to measure the functional status of patients with spinal disorders. It is comprised of 10 dimensions with 6 levels being set in each dimension.

SECONDARY OUTCOMES:
fear avoidance beliefs questionnaire (FABQ) | 5 minutes
  The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale, where 0= completely disagree, 6=completely agree.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No